CLINICAL TRIAL: NCT01187706
Title: A Controlled Study of Quality of Life and it's Related Factors Among Gynecological Cancer Survivors
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: National Taiwan University Hospital (Other)
Responsible Party: Fei-Hsiu Hsiao, National Taiwan University Hospital
Other Study IDs: 201007087R
Record Dates: First submitted 2010-08-23; First posted 2010-08-24 (Estimated); Last update posted 2010-08-24 (Estimated); Status verified 2010-08

CONDITIONS: Cervical Cancer; Ovarian Cancer; Endometrial Cancer
Keywords: gynecological cancer survivors; quality of life
MeSH Terms: conditions — Uterine Cervical Neoplasms; Ovarian Neoplasms; Endometrial Neoplasms

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- gynecological cancer survivors: Criteria for including: (1)Been diagnosed as cervical cancer, ovarian cancer or endometrial cancer, and has completed six months after the relevant treatment. (2)Age from 20 - 70 years old. (3) Agreed to participate in this study.
  Criteria for exclusion: Combined with other non-gynecologic cancer (cervical cancer, ovarian cancer or endometrial cancer) patients.
- healthy controls: Criteria for including: (1)Not those who suffer from cancer.(2)20-70 years old.(3)Agreed to participate in this study.Criteria for exclusion:Had undergone gynecologic surgical removal of ovaries or uterus were.

SUMMARY:
To compare quality of life and it's related factors between gynecological cancer survivor and healthy controls.

DETAILED DESCRIPTION:
This study used a cross-sectional design. By using the method of purposive sampling, the 70 gynecological cancer patients who had completed the active treatments for six months will be recruited from the oncology and gynecology clinics of a medical center in the Northern Taiwan area. The 70 healthy controls without any cancer will be recruited from clinic and from friends and colleagues. The instruments include "Sample characteristics questionnaire," "Short Form-12 (SF-12)," "Medical Outcome Study Sleep Scale (MOS-sleep)," "Beck Depression Inventory-II (BDI)," "State-Trait Anxiety Inventory (STAI)," "Sexual Activity Questionnaire (SAQ), and "The Experiences in Close Relationships-Revised (ECR-R)." The data will be analyzed by descriptive statistical analysis, independent t-test, ANOVA, Scheffe's test, Pearson's correlation, and stepwise regression.

ELIGIBILITY:
Inclusion Criteria:

* Been diagnosed as cervical cancer, ovarian cancer or endometrial cancer, and has completed six months after the relevant treatment.
* 20-70 years old
* Agreed to participate in this study.

Exclusion Criteria:

* Combined with other non-gynecologic cancer (cervical cancer, ovarian cancer or endometrial cancer) patients.

Ages: 20 Years to 70 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: This study used a cross-sectional design. By using the method of purposive sampling, the 70 gynecological cancer patients who had completed the active treatments for six months will be recruited from the oncology and gynecology clinics of a medical center in the Northern Taiwan area. The 70 healthy controls without any cancer will be recruited from clinic and from friends and colleagues.
Sampling Method: Non-Probability Sample
Enrollment: 140 (Estimated)
Dates: Start 2010-08

CONTACTS AND LOCATIONS:
Overall Officials: Fei-Hsiu Hsiao, Ph.D, Principal Investigator — National Taiwan University Hospital
Locations (1):
- National Taiwan University Hospital, Taipei, Taiwan